CLINICAL TRIAL: NCT01162486
Title: Phase I Dose Escalation Study of the Pharmacokinetics, Safety and Tolerability of Rifapentine and the Effects of Increasing Doses of Rifapentine on Induction of Metabolizing Enzymes in Healthy Volunteers
Brief Title: Pharmacokinetics, Safety and Tolerability of Escalating Rifapentine Doses in Healthy Volunteers
Acronym: TBTC S29B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Sanofi (Industry); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCHHSTP-5779
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-01

CONDITIONS: Tuberculosis; Tuberculosis, Pulmonary
Keywords: Anti-infective agents; Anti-bacterial agents; Rifampin; Rifapentine; Midazolam; Molecular mechanisms of pharmacological action; Antitubercular agents; Pharmacologic actions
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Pulmonary | interventions — Rifampin; Midazolam; rifapentine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Rifampin control (Active Comparator): Rifampin + midazolam
  Interventions: Drug: Rifampin & midazolam
- RPT 1 (Experimental): RPT Cohort 1 - 5 mg/kg
  Interventions: Drug: rifapentine & midazolam
- RPT 2 (Experimental): RPT Cohort 2 - 10 mg/kg
  Interventions: Drug: rifapentine & midazolam
- RPT 3 (Experimental): RPT Cohort 3 - 15 mg/kg
  Interventions: Drug: rifapentine & midazolam
- RPT 4 (Experimental): RPT Cohort 4 - 20 mg/kg
  Interventions: Drug: rifapentine and midazolam
- RPT 5 (Experimental): RPT Cohort 5 - Maximal tolerated dose, if dose limiting toxicities are observed
  Interventions: Drug: rifapentine and midazolam

INTERVENTIONS:
Drug: Rifampin & midazolam — rifampin - tablet, 10 mg/kg, daily 15 days midazolam - liquid syrup, 15 mg, days 1 and 15
  Arms: Rifampin control
Drug: rifapentine & midazolam — rifapentine - tablet, 5 mg/kg, daily 15 days midazolam - liquid syrup, 15 mg, days 1 and 15
  Arms: RPT 1
Drug: rifapentine & midazolam — rifapentine - tablet, 10 mg/kg, daily 15 days midazolam - liquid syrup, 15 mg, days 1 and 15
  Arms: RPT 2
Drug: rifapentine & midazolam — rifapentine - tablet, 15 mg/kg, daily 15 days midazolam - liquid syrup, 15 mg, days 1 and 15
  Arms: RPT 3
Drug: rifapentine and midazolam — rifapentine - tablet, 20 mg/kg, daily 15 days midazolam - liquid syrup, 15 mg, days 1 and 15
  Arms: RPT 4
Drug: rifapentine and midazolam — rifapentine - tablet, 2.5 mg/kg lower than previously tolerated dose cohort, daily 15 days midazolam - liquid syrup, 15 mg, days 1 and 15
  Arms: RPT 5

SUMMARY:
The aim of this study is to evaluate (1) the safety and tolerability of escalating doses of rifapentine (RPT) administered daily by oral; (2) the effect of increasing doses of RPT on cytochrome P450 isoform 3A (CYP3A) enzyme metabolizing activity, using single-dose midazolam (MDZ); and (3) the effect of increasing doses of RPT on autoinduction of RPT metabolism.

DETAILED DESCRIPTION:
On day 1, volunteers will receive a single dose of MDZ dosed at 15 mg delivered orally, and a 24-hour PK analysis of MDZ and its metabolite, 1-OH-midazolam (1-OH-MDZ) will be performed. RPT (or RIF) will be given as a single daily dose (5, 10, 15, or 20 mg/kg, depending on the dose cohort) on days 2-15 (14 doses). A 24-hour PK analysis of RPT (or RIF) and its 25-deacetyl metabolite (25-des-RPT) will be performed after the first dose (day 2). On day 15, volunteers receive a second single dose of MDZ. A 72-hour RPT (or RIF) and 24-hour MDZ (and 1-OH-MDZ) PK analysis will be performed after the second dose of MDZ beginning on day 15. The PK sampling will occur both on an in-patient basis in the General Clinical Research Center (GCRC) and on an out-patient basis in the study clinic. Volunteers will undergo assessments for adverse events (AEs) several times throughout the study.

Each dose cohort will contain 6 subjects. RPT dosing will begin at 5 mg/kg (6 volunteers) and increase by 5 mg/kg increments (6 volunteers each at 10, 15, and 20 mg/kg) to a maximum dose of 20 mg/kg unless dose-limiting toxicities (DLT) are seen in two or more patients within a dose cohort, in which case a dose that is 2.5 mg/kg lower than the previous dose will be enrolled to determine the maximal tolerated dose (MTD). In addition, one cohort of 6 subjects will receive RIF at 10 mg/kg daily, rather than RPT, as a comparator arm.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to provide written informed consent.
2. Age greater than or equal to 18 years, and less than or equal to 65 years.
3. Weight of 50-100 kg for enrollment into the RPT cohorts
4. Weight of 50-80 kg for enrollment into the RIF cohort
5. Within 28 or fewer days prior to enrollment, a complete blood count with differential, comprehensive serum chemistry profile, HIV antibody test, and Hepatitis C antibody test will be performed, with the following laboratory values:

   1. Serum amino aspartate transferase (AST) less than the upper limit of normal
   2. Total bilirubin level less than the upper limit of normal
   3. Serum creatinine <1.5 mg/dL
   4. Hemoglobin greater than 12.0 for men, greater than 11.0 for women
   5. Platelet count greater than or equal to 125,000 /cu mm
   6. Absolute neutrophil count greater than or equal to 1250 /cu mm
   7. Serum albumin greater than 3.5 g/dL
   8. HIV antibody test negative
   9. Hepatitis C antibody negative
6. For women of childbearing potential, a negative serum bHCG pregnancy test, performed at screening.
7. During the study and for 14 days after the last dose of study medication, women of childbearing potential must agree to practice barrier contraception for the duration of the study.

Exclusion Criteria:

1. Pregnant or breastfeeding
2. Known intolerance of or allergy to rifamycins
3. Allergy to benzodiazepines
4. Use of rifamycin antibiotics in the 30 days prior to enrollment
5. Inability to take oral medications
6. Renal, hepatic, cardiac (except benign heart murmur), or endocrine disorder; or malignancy; or immunocompromise.
7. History of any acute or chronic illness that requires current medical therapy.
8. Prior gastrointestinal surgery involving stomach, biliary system, pancreas, or small intestine.
9. Any medical condition that, in the opinion of the investigator, would interfere with the subject's ability to participate in the protocol.
10. Any illicit drug use within the preceding 2 months. Subjects must agree to abstain from alcohol and illicit drug use during the study. Smokers must agree to abstain from cigarettes or to smoke fewer than 5 cigarettes per day.
11. Current use of any prescription medication(s), including oral contraceptives.
12. Planned use, during the study from Day 0 through the last PK blood draw, of any of the following: prescription medication(s), herbal supplement(s), vitamin(s), mineral supplement(s), over-the-counter medication(s), or grapefruit juice. Subjects must agree to abstain from grapefruit juice during the study.
13. Participation in any other investigational drug study within 30 days prior to study entry and during study.
14. Inability to participate in pharmacokinetic visits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Dooley, MD, PhD, Principal Investigator — Johns Hopkins University; Susan Dorman, MD, Principal Investigator — Johns Hopkins Univeristy
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Savic RM, Lu Y, Bliven-Sizemore E, Weiner M, Nuermberger E, Burman W, Dorman SE, Dooley KE. Population pharmacokinetics of rifapentine and desacetyl rifapentine in healthy volunteers: nonlinearities in clearance and bioavailability. Antimicrob Agents Chemother. 2014 Jun;58(6):3035-42. doi: 10.1128/AAC.01918-13. Epub 2014 Mar 10. PMID 24614383

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rifampin Control | RPT 1 | RPT 2 | RPT 3 | RPT 4
Started | 8 | 6 | 6 | 7 | 6
Took at Least One Dose Study Drug | 8 | 6 | 6 | 7 | 6
Completed | 6 | 6 | 5 | 6 | 6
Not Completed | 2 | 0 | 1 | 1 | 0
Not completed — low ANC | 1 | 0 | 0 | 0 | 0
Not completed — vomited Rifampin/ gagged with midazolam | 1 | 0 | 0 | 0 | 0
Not completed — elevated LFTs | 0 | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: 4 of the enrolled participants did not get to start. Two withdrew their consent, one had a transaminase elevation and one was non-compliant. Only 33 (out of the 37 enrolled participants) were able to start the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rifampin Control | RPT 1 | RPT 2 | RPT 3 | RPT 4 | Total
Number analyzed (Participants) | 8 | 7 | 7 | 7 | 8 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 7 | 7 | 8 | 37
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 39 [25 to 50] | 50 [29 to 55] | 44 [27 to 58] | 41 [23 to 59] | 47 [30 to 55] | 44 [23 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 3 | 1 | 6
  Male | 7 | 6 | 7 | 4 | 7 | 31
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 7 | 7 | 8 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 2 or Higher Adverse Events Over the Course of the 26 Day Trial
Description: Number of Participants with Grade 2 or higher adverse events over 26 days
Time Frame: 26 days
Population: Four withdrew prior to receiving study rifamycin so were not included in the safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Rifampin Control | RPT 1 | RPT 2 | RPT 3 | RPT 4
Number analyzed (Participants) | 8 | 6 | 6 | 7 | 6
Participants | 1 | 0 | 1 | 1 | 0

2. Primary Outcome: Pharmacokinetics (AUC of RPT Over 24 Hours Post-dose)
Description: To determine and compare the steady-state pharmacokinetics and dose linearity of escalating daily doses of rifapentine in dose cohorts of 5 mg/kg, 10 mg/kg, 15 mg/kg and 20 mg/kg in healthy volunteers after a single dose (Day 2) or multiple doses (Day 15)
Time Frame: days: 2, 15
Population: These patients completed PK visits on Day 2 and 15 (Three participants in this non-control group - subdivided into 4- did not complete the study). Reasons provided in the participant flow session
Measure: Median (Full Range); unit: (mcg*h/ml)
Arm/Group | RPT 1 | RPT 2 | RPT 3 | RPT 4
Number analyzed (Participants) | 5 | 5 | 6 | 6
(mcg*h/ml)
  RPT AUC, Day 2 single dose | 128 [101 to 157] | 242 [231 to 260] | 363 [310 to 430] | 403 [357 to 452]
  RPT AUC, Day 15 multiple dose | 218 [142 to 251] | 330 [284 to 340] | 560 [401 to 735] | 483 [414 to 546]

3. Secondary Outcome: Midazolam, AUC Over 12 Hours Post-dose
Description: To compare and describe, the pharmacokinetics of single-dose midazolam alone (Day 1) versus midazolam co-administered with either steady-state rifapentine at multiple daily doses (5, 10, 15, and 20 mg/kg) or rifampin at 10 mg/kg daily (Day 15)
Time Frame: days: 1, 15
Population: 29 participants completed both midazolam PK visits; one person in RPT1 visit was not analyzed because his samples were zero and was found to have been non-compliant with regimen
Measure: Median (Full Range); unit: ng*h/ml
Arm/Group | Rifampin Control | RPT 1 | RPT 2 | RPT 3 | RPT 4
Number analyzed (Participants) | 6 | 5 | 5 | 6 | 6
ng*h/ml
  AUC 0-12 Midazolam alone (Day 1) | 151 [116 to 197] | 150 [108 to 238] | 114 [111 to 128] | 204 [158 to 255] | 173 [118 to 270]
  AUC 0-12 Midazolam with RIF (Day 15) | 26.9 [10.0 to 55.8] | 14.2 [7.34 to 20.1] | 10.2 [10.0 to 10.4] | 14.0 [12.6 to 15.2] | 11.7 [8.8 to 14.6]

4. Secondary Outcome: Transporter Genes
Description: To determine the effects of polymorphisms of transporter genes on rifampin and rifapentine PK parameters
Time Frame: day 3
Population: This outcome was not assessed because data was not collected
Arm/Group | Rifampin Control | RPT 1 | RPT 2 | RPT 3 | RPT 4
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Rifapentine Concentrations From Dried Blood Spots
Description: To develop methods for determination of rifapentine concentrations from dried blood spots on sampling paper
Time Frame: days 2, 3, 7, 10, 15, 16, 17, 18
Population: This outcome was not assessed because data was not collected
Arm/Group | Rifampin Control | RPT 1 | RPT 2 | RPT 3 | RPT 4
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Rifampin Control | RPT 1 | RPT 2 | RPT 3 | RPT 4
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 5/8 | 2/6 | 3/6 | 4/7 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rifampin Control (N=8) | RPT 1 (N=6) | RPT 2 (N=6) | RPT 3 (N=7) | RPT 4 (N=6)
Gas (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Vomitting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lymphopenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperglycemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasemia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No